CLINICAL TRIAL: NCT05871502
Title: Glycemia and Ischemia Reperfusion Brain Injury in Patients With Acute Cerebral Infarction Treated With Mechanical Thrombectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GLIAS-TM
Record Dates: First submitted 2023-04-14; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Intervention Model Description: Before the start of the endovascular procedure, a subcutaneous blood glucose monitoring device will be implanted, which will be removed on day 15 (or at hospital discharge if this takes place before 15 days). Those patients with blood glucose levels >155 mg/dl will receive insulin at the discretion of the physician responsible for the patient, following the local protocols for the management of hyperglycemia in hospitalized patients and the guidelines for the management of hyperglycemia in patients with acute stroke.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subcutaneous blood glucose monitoring device (Experimental): After signing the informed consent and before the start of the endovascular procedure, a subcutaneous blood glucose monitoring device will be implanted, which will be removed on day 15 (or at hospital discharge if this takes place before 15 days).
  Interventions: Device: Subcutaneous blood glucose monitoring device

INTERVENTIONS:
Device: Subcutaneous blood glucose monitoring device — After signing the informed consent and before the start of the endovascular procedure, a subcutaneous blood glucose monitoring device will be implanted, which will be removed on day 15 (or at hospital discharge if this takes place before 15 days). This device will be selected from those currently available on the market, with CE marking, and with previous studies documenting its safety and feasibility for radiological procedures.

SUMMARY:
Postictus hyperglycemia is associated with an accelerated transformation of the ischemic penumbra into an infarct area, with increased infarct size, worse recanalization, reduced cerebral perfusion, increased ischemia reperfusion damage, and worse outcome. Furthermore, when perfusion is reinstated, hyperglycemia causes secondary tissue damage through an increase in ischemic reperfusion damage. Thus, those patients with glycemia values < 155 mg/dL during mechanical thrombectomy, and especially at the time of reperfusion, will have greater ischemia-reperfusion damage, showing a different profile in miRNA expression, with better neurological and functional outcomes and higher risk of hemorrhagic transformation and cerebral edema.

The main objective of the study is to evaluate the association between glycemia values at the time of reperfusion and stroke recovery at 3 months in patients with acute cerebral infarction treated with mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Neuroimaging studies such as computed tomography (CT), angio-CT or angio-MRI compatible with the diagnosis of acute cerebral infarction due to occlusion of a large vessel of the anterior circulation, including the internal carotid artery (intra- or extracranial) or middle cerebral artery (M1 or M2 segments).
* Indication of mechanical thrombectomy according to clinical practice.
* Inclusion of the patient in the study before the endovascular procedure.
* Modified Rankin Scale (mRS) score prior to stroke of 0-1.
* Signature of informed consent.

Exclusion Criteria:

* CT, angio-CT or angio-MRI showing posterior circulation occlusion.
* Severe or life-threatening concomitant disease that precludes follow-up for 3 months after stroke,
* Alcohol or drug abuse
* Participation in a therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-04-13 (Estimated); Study Completion 2025-04-13 (Estimated)

PRIMARY OUTCOMES:
Blood glucose levels at the time of reperfusion | During reperfusion procedure
  Blood glucose levels at the time of reperfusion in patients achieving TICI-2b, TICI-2c or TICI3 recanalization pattern after mechanical thrombectomy.
Modified Rankin scale at 3 months | From baseline to month 3
  Its dichotomized assessment (Modified Rankin Scale or mRS 0-2 indicating good functional recovery and 3-6 indicating death or dependence) is commonly used in acute stroke studies.

SECONDARY OUTCOMES:
Peak blood glucose values | During the mechanical thrombectomy procedure
  Peak blood glucose values during the mechanical thrombectomy procedure.
Blood glucose values above 155 mg/dL | The entire time from arrival at the emergency room until completion of the arterial recanalization procedure.
  Total time with blood glucose values above 155 mg/dL from arrival at the emergency department to arterial recanalization
Time in range 110-154 mg/dL of blood glucose values | From arrival at the emergency department to recanalization, during the first 24 hours and during hospital stay
  Time in range 110-154 mg/dL of blood glucose values: (a) from arrival at the emergency department to recanalization; (b) during the first 24 h; and (c) during hospital stay
Proportion of patients receiving insulin treatment | During the first 24 hours from the onset of stroke symptoms
  Proportion of patients receiving insulin treatment for post-stroke hyperglycemia, during the first 24h from the onset of stroke symptoms
Dose of insulin treatment received by clinical practice | Through study completion, an average of 2 years
  Insulin treatment received by clinical practice (route of administration and dose)
Number of subcutaneous blood glucose monitoring devices with technical failures | Through study completion, an average of 2 years
  Number of subcutaneous blood glucose monitoring devices with technical failures (absence or interruption of readings) or requiring replacement due to involuntary removal of the device or inadequate implantation.
Additional data of the subcutaneous blood glucose monitoring device | During the time the device is worn, up to 15 days
  Mean blood glucose
Number of mechanical thrombectomy passes | Through study completion, an average of 2 years
  Number of mechanical thrombectomy passes (includes aspirations and stent-retriever passes).
Degree of recanalization | Through study completion, an average of 2 years
  Degree of recanalization according to the TICI classification in the final angiogram (from no perfusion (grade 0) to complete perfusion (grade 3))
Arterial blood pressure | During reperfusion procedure
  Arterial blood pressure in the emergencies and at the time of reperfusion.
Infarct size | At 24 hours
  Infarct size at 24 hours (assessed by a radiologist who will be unaware of blood glucose monitoring data)
Hemorrhagic transformation | At 24 hours
  Hemorrhagic transformation at 24 hours (assessed by a radiologist who will be unaware of blood glucose monitoring data). It will be categorized into four types: (1) hemorrhagic infarction type 1 (HI-1): small petechiae at the edges of the infarcted area; (2) hemorrhagic infarction type 2 (HI-2): confluent petechiae in the infarct area without mass effect; (3) parenchymal hematoma type 1 (HP-1): hematoma occupying ≤ 30% of the infarct area, with discrete mass effect; and (4) parenchymal hematoma type 2 (HP-2): hematoma occupying more than 30% of the infarct area, with evident mass effect.
Number of symptomatic hemorrhagic transformation | During a symptomatic hemorrhagic transformation
  Symptomatic hemorrhagic transformation defined as computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of any type of hemorrhage that is accompanied by neurological deterioration ≥ 4 points on the National Institutes of Healt Stroke Scale scale from baseline or leading to death.
National Institutes of Healt Stroke Scale score | At 24 hours and at 3 months
  National Institutes of Healt Stroke Scale score at 24 hours, at hospital discharge, and at 3 months (scores range from 0 to 42, with higher scores indicating more severe neurological deficit).
Neurological or systemic complications | During follow-up period, up to 3 months
  Neurological or systemic complications during follow-up. The following complications will be systematically assessed at each visit: coma, seizures, early neurological deterioration, cerebral edema, recurrent stroke, acute coronary syndrome, pulmonary thromboembolism, respiratory infection, urinary tract infection, sepsis, local hematoma or infection at the insertion site of the subcutaneous blood glucose monitor. Any other complication that is referred or detected during follow-up will also be recorded.
Distribution of scores on the modified Rankin scale | At 90 days
  Distribution of scores on the modified Rankin scale at 90 days (shift analysis).
Mortality | At 3 months
  Mortality at 3 months
Presence of biomarkers of ischemia-reperfusion injury | During reperfusion procedure and 24 hours later
  Biomarkers of ischemia-reperfusion injury: miR-29b, miR-339, miR-15a, miR-100 and miR-424. Samples will be collected at the time of reperfusion and 24 hours later.

OTHER OUTCOMES:
Demographic data: | Through study completion, an average of 2 years
  Age, sex, race, weight, height, previous diagnosis or treatment for any of the following conditions: diabetes, hypertension, dyslipidemia, coronary artery disease, atrial fibrillation, metabolic syndrome, chronic kidney disease (eGFR < 60 ml/min/1.73m2), smoking or alcohol abuse.
Number of previous pharmacological treatments | Before entering the study
  Platelet antiaggregants, anticoagulants, antihypertensives, antidiabetics and lipid-lowering agents.
Stroke data | During the duration of the stroke
  Date of symptom onset (or last asymptomatic in patients with unknown stroke onset), subtype of stroke and treatment with intravenous thrombolysis.
Neuroimaging data | At the baseline visit
  Baseline ASPECTS (degree of collateral circulation and perfusion)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hervas C, Peiroten I, Gonzalez L, Alonso de Lecinana M, Alonso-Lopez E, Casado L, De Celis-Ruiz E, Fernandez Prieto AF, Frutos R, Gallego-Ruiz R, Gonzalez Perez de Villar N, Gutierrez-Fernandez M, Navia P, Otero-Ortega L, Pozo-Novoa J, Rigual R, Rodriguez-Pardo J, Ruiz G, Fuentes B. Glycaemia and ischaemia-reperfusion brain injury in patients with ischaemic stroke treated with mechanical thrombectomy (GLIAS-MT): an observational, unicentric, prospective study protocol. BMJ Open. 2024 Aug 7;14(8):e086745. doi: 10.1136/bmjopen-2024-086745. PMID 39117402